CLINICAL TRIAL: NCT00714025
Title: A Single Arm, Multicenter, Phase II Trial of RAD001 as Monotherapy in the Palliative Treatment of Patients With Locally Advanced or Metastatic Transitional Cell Carcinoma After Failure of Platinum-based Chemotherapy
Brief Title: A Single Arm, Multicenter, Phase II Trial of RAD001 as Monotherapy in the Palliative Treatment of Patients With TCC After Failure of Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL-ONCO 08-002
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Transitional Cell Carcinoma
Keywords: RAD001; TCC; Palliative treatment; advance or metastatic TCC; Failure after Platinum-based chemotherapy
MeSH Terms: conditions — Carcinoma, Transitional Cell; NOG-Related-Symphalangism Spectrum Disorder | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): 40 patients with metastatic or locally advanced transitional bladder cancer with failed platinum-based chemotherapy receiving RAD001 10mg daily PO.
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — RAD001 10mg, daily, PO

SUMMARY:
An open-label, single arm, non-randomized, single stage phase II study. 3 phases:Baseline, treatment/duration and Follow-up. All patients will be treated with RAD001 10 mg daily dose until disease progression or unacceptable toxicity death, or discontinuation from the study, for any other reason

DETAILED DESCRIPTION:
An open-label, single arm, non-randomized, single stage phase II study. Baseline phase: Baseline evaluations will be performed within 2 weeks before the first dose study drug.

Treatment phase/duration of treatment: All patients will be treated with RAD001 10mg PO daily dose until disease progression (by RECIST) or unacceptable toxicity death or discontinuation from the study for any other reason.

Follow-up phase: All patients will have a follow-up visit scheduled 28 days after the last dose of the study drug to follow for AEs and SAEs that may have occured after discontinuation from the study. Any patient who is discontinued from treatment with RAD001 for any reason other than disease progression will continue to have tumor assessments until the patient has documented disease progression or start of additional anti-tumor therapy. Central radiology review and survival data collection will be performed. After discontinuation of RAD001 all patients will be followed up for survival until the final OS analysis is performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients histologically-or cytologically-confirmed locally advanced or metastatic TCC not amenable to curative surgery or radiation.
* Patients with documented disease progression after first-line platinum based therapy
* an interval of more than 4 weeks since last cytotoxic chemotherapy, biological therapy, surgery or radiotherapy
* patients with at least one measurable lesion as at baseline as per RECIST criteria
* ECOG performance status of 0-2
* Adequate bone marrow function
* Adequate liver function
* Adequate renal function
* Life expectancy more than 3 months
* Women of child-bearing age must have a negative pregnancy test within 72 hours prior to the administration of the study treatment start
* Signed informed consent prior to beginning protocol specific procedure
* Age more than 18 years old

Exclusion Criteria:

* Patients who have received more than 2 systemic treatment for their metastatic disease
* Patients who have previously received mTOR inhibitors
* Patients with a know hypersensitivity to RAD001 or other rapamycin or to its recipients
* Patients with brain or leptomeningeal metastases
* Patients receiving chronic systemic treatment with corticosteroids or another immunosuppressive agent
* Patients with a known history of HIV seropositivity
* Patients with autoimmune hepatitis
* patients with an active, bleeding diathesis
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Patients who have a history of another primary malignancy more than 5 years
* Patients who are using other investigational agents or who had received investigational drugs more than 4 weeks prior to study treatment start
* Patients unwilling to or unable to comply with the protocol
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Oral contraceptives are not acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Primary:To evaluate the preliminary efficacy of RAD001 as monotherapy for the treatment of locally advanced or metastatic TCC. Efficacy is defined as the disease control rate at 8 weeks. | 8 weeks

SECONDARY OUTCOMES:
Secondary:To evaluate the response rate, duration of response, progression-free survival and overall survival in this patient population, and further characterize the safety profile of RAD001 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal H Machiels, MD PhD, Principal Investigator — Cliniques Universitaires St Luc-UCL
Locations (1):
- Cliniques Universitaires St Luc-UCL, Brussels, Belgium